CLINICAL TRIAL: NCT03097809
Title: SEEG Investigation of Mood Dysregulation in People With Epilepsy
Brief Title: SEEG Investigation of Mood Dysregulation in Epilepsy
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Amit Anand, MD, MD, The Cleveland Clinic
Other Study IDs: 15-1007
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epilepsy Subjects: Subjects will be recruited from the epilepsy-monitoring unit. These subjects would have been already assessed by the Epilepsy Center at the Cleveland Clinic for surgical treatment of medically refractory epilepsy and would have already had SEEG electrodes placed in cortical and limbic areas for clinical diagnostic purposes.
  Interventions: Other: SEEG Recordings

INTERVENTIONS:
Other: SEEG Recordings — To directly record brain activity from the frontal-limbic circuitry of subjects in the resting state and while they engage in behavioral tasks designed to assess emotional response to negative stimuli and different aspects of impulse control and emotional processing

SUMMARY:
Using the novel analysis of stereo-electroencephalography (SEEG) recordings, this proposal will investigate the activity and connectivity of mood regulation circuits in subjects with suspected epileptic focus who have undergone SEEG electrode implantation for monitoring of seizure activity.

DETAILED DESCRIPTION:
It is well known that epilepsy is associated with mood dysregulation including symptoms of labile mood, impulse control problems, anxiety, depression and increase in incidence of suicide. However, until present the neurobiological basis of mood dysregulation in epilepsy has not been clear and has been mostly attributed to a psychological reaction to the illness. This has severely limited our understanding of the impairments in mood regulation that people with epilepsy often experience and has also limited the development of effective treatment for ameliorating psychosocial dysfunction in people with epilepsy. The identification of these circuits will not only increase our understanding of mood-regulation in epilepsy but also possibly provide biomarkers with which the effectiveness of new treatments can be investigated. Developing better diagnostic measures and treatments for mood dysregulation will be highly beneficial to the quality of life of subjects suffering from epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be a part of the epilepsy-monitoring unit for long-term SEEG recordings and analysis

Exclusion Criteria:

* Subjects that experience surgical complications during the implant procedure will be excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects from the Epilepsy Center at the Cleveland Clinic for surgical treatment of medically refractory epilepsy who would have already had SEEG electrodes placed in cortical and limbic areas for clinical diagnostic purposes
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Emotional Face Task and Emotional Go-No Go Task | 2 years
  To use face pictures depicting negative, positive and neutral emotions this task measures brain area activation abnormalities while responding and inhibiting responses to positive and negative emotions.
Maintaining and suppressing emotions | 2 years
  To use the International Affective Picture System, subjects will be asked to either maintain or suppress their emotions.
Resting state cortico-limbic brain connectivity | 2 years
  Resting state recordings will be collected from the cortical areas - prefrontal cortex, orbitofrontal cortex and anterior and posterior cingulate cortex as well as limbic areas - amygdala and hippocampus

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation Center for Behavioral Health, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No